CLINICAL TRIAL: NCT05737316
Title: A Randomised Controlled Feasibility Study of a Novel Technology-assisted Home Based Aerobic Exercise Programme for Individuals With Parkinson's Disease
Brief Title: A Novel Technology-assisted Home Based Aerobic Exercise Programme for Individuals With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Singhealth Foundation (Other Government)
Responsible Party: Principal Investigator, Chloe Chung Lau Ha, Principal Physiotherapist, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/00768
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: exercise; Gamification
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient blinding will be done by ensuring that patients are unaware of the content of either treatment group before participation, and will only be made aware of the content of their allocated programme after randomization. They will be instructed not to share the details of their exercise programme with their physicians or other study participants, and to only contact their assigned physiotherapist in case of any problems during the study. Intervention and control group participants will be assigned different dates for study site visits to avoid cross-contamination.
  Study team members who will assess outcomes or perform data analyses will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combat PD (Experimental): Combat PD is an aerobic exercise programme hosted on a mobile application.
  Interventions: Behavioral: Combat PD
- Usual Care (Active Comparator): Home exercises based on a standard PD exercise booklet, consisting mainly of range of motion and stretching exercises
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Combat PD — CombatPD is an aerobic exercise programme hosted on a mobile application that pairs with motion sensors and heart rate monitor, which connects to a web-based portal for remote monitoring. The wearable sensors consist of (i) 2 motion sensors worn across one thigh and attached to an exercise ring which is held by the participant during the exergame and (ii) 1 heart rate sensor worn across the participant's chest. They will receive once weekly physiotherapy sessions at the study site for the first 4 weeks where they will be guided through the use of the CombatPD. Participants will be instructed to perform 2 sessions of 30-minute exergames in addition to a session of 30-minute brisk walking every week for 12 weeks at home. They will be instructed to exercise at a target heart rate zone at moderate intensity (i.e., 40% - 60% Heart Rate Reserve), which will be gradually increased.
  Arms: Combat PD
Behavioral: Usual Care — Participants in the control group (usual care) will receive once weekly physiotherapy sessions for first 2 weeks and another session at week 6 where they will be taught home exercises based on a standard PD exercise booklet, consisting mainly of range of motion and stretching exercises , as well as brisk walking techniques. Participants in the control group will be instructed to perform these home exercises twice a week, in addition to a 30-minute brisk walk for 12 weeks.
  Arms: Usual Care

SUMMARY:
This study aim to evaluate the (1) feasibility of a novel mobile application ( Combat PD) that support a home-based gamified aerobic exercise program in individuals with mild Parkinson's disease (PD).

The study aims to further explore (2) the effectiveness of Combat PD in improving adherence to prescribed home-based exercise program; and (3) the clinical effectiveness if combat PD in improving motor and non-motor function in PD.

DETAILED DESCRIPTION:
This study aim to evaluate the (1) feasibility of a novel mobile application ( Combat PD) that support a home-based gamified aerobic exercise program in individuals with mild Parkinson's disease (PD).

The study aims to further explore (2) the effectiveness of Combat PD in improving adherence to prescribed home-based exercise program; and (3) the clinical effectiveness if combat PD in improving motor and non-motor function in PD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 30-75, diagnosed with Parkinson's disease, with mild disease severity (Hoehn and Yahr stages I to II)
2. Sedentary lifestyle
3. Receive a stable dose of dopaminergic medication for at least 4 weeks prior to study inclusion
4. Has a smart phone device

Exclusion Criteria:

1. Uncontrolled hypertension, arrhythmia, or unstable cardiovascular status
2. Poorly controlled diabetes mellitus
3. Advanced kidney disease
4. BMI > 30
5. Recent cerebrovascular event/ concussion/ fall in the last 6 months
6. Significant cognitive impairment (MoCA<21)
7. Any other medical/orthopaedic/psychiatric condition that would interfere with ability to participate in the study
8. No stable internet or smart device access
9. Inability to fill up self-reported questionnaires
10. Attendance at any regular exercise programme up to 4 weeks prior to study inclusion

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-11 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to exercise program | 12 weeks
  actual exercise frequency compared to prescribed exercise targets.
Adherence to exercise program | 12 weeks
  actual exercise duration compared to prescribed exercise targets.
Adherence to exercise program | 12 weeks
  actual exercise intensity (period of exercise performed within prescribed heart rate zone), compared to prescribed exercise targets.

SECONDARY OUTCOMES:
Adverse events | 12 weeks
  Falls, musculoskeletal injuries, shortness of breath, dizziness, and fatigue.
Motor section of Movement Disorder Society sponsored Unified Parkinson's disease Rating Scale (MDS-UPDRS-III) | 12 weeks
  Motor section of Movement Disorder Society sponsored Unified Parkinson's disease Rating Scale (MDS-UPDRS-III) is a valid and reliable clinical test to evaluate the severity of motor symptoms of PD, score range 0-132, 32 and below is mild, 59 and above is severe.
Timed Up and Go test (TUG) | 12 weeks
  The TUG test measures the time in seconds taken by participants to perform sequential locomotor tasks that incorporate walking and turning.
Dual-task Timed Up and Go Test (TUG) | 12 weeks
  Participants were instructed to repeat the TUG procedure while performing a serial three subtraction.
6-minute walk test | 12 weeks
  The maximal distance covered over a time of 6 minute.
Montreal Cognitive Assessment (MoCA) | 12 weeks
  MoCA is a widely used screening assessment for detecting cognitive impairment, The basics of this test include short-term memory, executable performance, attention, focus and more. Score range 0-30. A score of 26 or over is considered to be normal.
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  A reliable instrument for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic. The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from 0 to 3, with 3 denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Fatigue Severity Scale (FSS) | 12 weeks
  The 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Score range from 9-63, higher the score denotes greater fatigue severity.
Scales for Outcomes in Parkinson's disease (SCOPA-sleep) | 12 weeks
  SCOPA-sleep is a reliable and valid patient-completed instrument for assessing nighttime sleep (5 items, 0-4) and daytime sleepiness (6 items 0-4) in patients with PD. with two additional questions on use of sleeping tablet ( 0-4) and Global evaluation of sleeping at night (0-7), sum up to total score of 55, higher score denotes worst sleeping performance.
Parkinson Disease Questionnaire (PDQ)-8 | 12 weeks
  It's a self-administered questionnaire, used to measure quality of life in persons with PD. It is an eight-question instrument and each score is scored between 0 and 4. Total score sum up to 32, a higher score signifies poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
individual participant data that underlie the results reported, after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 years after completion
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Background] Canning CG, Allen NE, Dean CM, Goh L, Fung VS. Home-based treadmill training for individuals with Parkinson's disease: a randomized controlled pilot trial. Clin Rehabil. 2012 Sep;26(9):817-26. doi: 10.1177/0269215511432652. Epub 2012 Jan 18. PMID 22257506
- [Background] van der Kolk NM, de Vries NM, Penko AL, van der Vlugt M, Mulder AA, Post B, Alberts JL, Bloem BR. A remotely supervised home-based aerobic exercise programme is feasible for patients with Parkinson's disease: results of a small randomised feasibility trial. J Neurol Neurosurg Psychiatry. 2018 Sep;89(9):1003-1005. doi: 10.1136/jnnp-2017-315728. Epub 2017 Jun 12. No abstract available. PMID 28607121